CLINICAL TRIAL: NCT00425061
Title: Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 2 Study Conducted Sequentially With 3 Doses Of Ima-638 Administered Sc.
Brief Title: Study Evaluating the Effect of IMA-638 in Subjects With Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3174K1-201; B2421007 (Other: Alias Study Number)
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — anrukinzumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Biological: IMA-638
- 2 (Experimental)
  Interventions: Biological: IMA-638
- 3 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Biological: IMA-638 — SC Injection, 12 weeks
  Arms: 1
Biological: IMA-638 — SC Injection, 12 weeks
  Arms: 2
Other: placebo — placebo
  Arms: 3

SUMMARY:
Primary purpose is to assess if IMA-638 is safe and improves asthma in subjects with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy men and women with persistent asthma, 18 to 70 years of age, with body weight between 50 kg and 115 kg.
* History of treatment with a medium to high dose of inhaled corticosteroids (ICS), with or without long-acting beta-agonists (LABA), for at least 2 months prior to the screening visit and must remain constant during the study.
* FEV1 ≥ 55% to ≤ 80% predicted and demonstrated improvement in FEV1 (L) with inhaled albuterol (salbutamol) (reversibility) of ≥ 12%.

Exclusion Criteria:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2007-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (82):
- United States (76):
  - Alabama Allergy and Asthma Center, Birmingham, Alabama
  - Alabama Allergy & Asthma Clinic, Montgomery, Alabama
  - Little Rock Allergy & Asthma, Little Rock, Arkansas
  - Pacific Coast Allergy, Crescent City, California
  - ABM Research Center, Fresno, California
  - Allergy and Asthma Care Center of Southern California, Long Beach, California
  - Allergy Medical Clinic, Los Angeles, California
  - Advances in Medicine, Rancho Mirage, California
  - Penisula Research Associates, Rolling Hills Estates, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Allergy Associates Medical Group, Inc., San Diego, California
  - Allergy & Asthma Assoc of Santa Clara Valley Research Ctr, San Jose, California
  - San Jose Clinical Research, Inc., San Jose, California
  - Bensch Research Associates, Stockton, California
  - Allergy and Immunology Medical Group, Vista, California
  - Allergy & Asthma Clinical Research, Inc., Walnut Creek, California
  - National Jewish Medical & Research Center, Denver, Colorado
  - Colorado Allergy and Asthma Centers, Denver, Colorado
  - Waterbury Pulmonary Associates, Waterbury, Connecticut
  - Brandon-Valico Center for Allergy & Asthma Research, LLC, Valrico, Florida
  - Roberson Allergy & Asthma, West Palm Beach, Florida
  - Georgia Pollens CRC, Inc., Albany, Georgia
  - DataQuest Medical Research, Lawrenceville, Georgia
  - Aero Allergy Research Labs of Savannah, Inc. 505 Eisenhower, Savannah, Georgia
  - Allergy and Asthma Center of Chicago, River Forest, Illinois
  - Fort Wayne Medical Institute, Fort Wayne, Indiana
  - South Bend Clinic, South Bend, Indiana
  - College Park Family Care Center, Overland Park, Kansas
  - Kansas City Allergy & Asthma, Overland Park, Kansas
  - Abraham Research, PLLC, Crescent Springs, Kentucky
  - Clinical Research Specialists, Metairie, Louisiana
  - Allergy and Arthritis Family, Gardner, Massachusetts
  - Center for Clinical Research, Taunton, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - Mississippi Asthma and Allergy Clinic, P.A., Jackson, Mississippi
  - Midwest Clinical Research LLC, St Louis, Missouri
  - The Clinical Research Center LLC, St Louis, Missouri
  - Montana Medical Research, Inc, Missoula, Montana
  - Midwest Allergy and Asthma Clinic, Omaha, Nebraska
  - Allergy and Asthma Assoc, Las Vegas, Nevada
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Pulmonary and Allergy Associates, Summit, New Jersey
  - Pulmonary & Critical Care Services, P.C.5 Palisades Dr., Su, Albany, New York
  - AAIR Research Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Regional Allergy and Asthma Consultants, P.A., Asheville, North Carolina
  - AAC Research, PC, Mt Pleasant, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Allergy & Respiratory Center, Canton, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Toledo Center for Clinial Researcch, Sylvania, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy and Asthma Research Group, Eugene, Oregon
  - Allergy, Asthma and Dermatology Research Center, LLC 3975 Me, Lake Oswego, Oregon
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Valley Clinical Research Center, Bethlehem, Pennsylvania
  - Allergy & Asthma Research of New Jersey, Philadelphia, Pennsylvania
  - Allergy and Clinical Immunology, Pittsburgh, Pennsylvania
  - Pulmonary and Allergy Associates, Sellersville, Pennsylvania
  - AAPRI Clinical Research Institute, Lincoln, Rhode Island
  - Allergic Disease and Asthma Center Research, PA, Greenville, South Carolina
  - AAC Research, PC, Mt. Pleasant, South Carolina
  - East Tennessee Center for Clinical Research, Knoxville, Tennessee
  - Lovelace Scientific Resources, Austin, Texas
  - Allergy and Asthma Research Center of El Paso, El Paso, Texas
  - Family Center for Asthma & Allergic Diseases, Friendswood, Texas
  - Allergy and Asthma Associates, Houston, Texas
  - Clinical Trials North Houston, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - The Allergy and Asthma Clinic of Central Texas, Killeen, Texas
  - Allergy Asthma and Immunology, San Antonio, Texas
  - Timber Lane Allergy and Asthma Research LLC, South Burlington, Vermont
  - Virginia Adult & Pediatric Allergy & Asthma, P.C., Richmond, Virginia
  - University of Wisconsin Medical School, Madison, Wisconsin
  - Auroroa Health Care, Inc., Milwaukee, Wisconsin
- Canada (6):
  - Alpha Medical Research Inc., Mississauga, Ontario
  - Alexander Medical Innovations Inc., Niagara Falls, Ontario
  - Allergy and Asthma Research Centre, Ottawa, Ontario
  - Recherche Invascor Inc, Longueuil, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CIC Mauricie Inc., Trois-Rivières, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3174K1-201&StudyName=Study%20Evaluating%20the%20Effect%20of%20IMA-638%20in%20Subjects%20With%20Persistent%20Asthma

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study had adaptive study design wherein participants were treated in 3 stages with higher number of participants enrolled in subsequent stages. As the treatment regimen was same for participants who received IMA-638 200 mg or placebo in Stage 2 and 3, participants were summarized together for these arms.
Groups:
- IMA-638 0.2 mg/kg: Stage 1: IMA-638 0.2 milligram/kilogram (mg/kg) subcutaneous injection on Day 1, 8, 28, 56 and 84 during Stage 1.
- IMA-638 0.6 mg/kg: Stage 1: IMA-638 0.6 mg/kg subcutaneous injection on Day 1, 8, 28, 56 and 84 during Stage 1.
- IMA-638 2 mg/kg: Stage-1: IMA-638 2 mg/kg subcutaneous injection on Day 1, 8, 28, 56 and 84 during Stage 1.
- Placebo: Stage 1: Placebo matched to IMA-638 subcutaneous injection on Day 1, 8, 28, 56 and 84 during Stage 1.
- IMA-638 200 mg: Stage 2 and 3: IMA-638 200 milligram subcutaneous injection on Day 1, 8, 28, 42, 56, 70 and 84 during Stage 2 and 3.
- IMA-638 75 mg: Stage 3: IMA-638 75 milligram subcutaneous injection on Day 1, 8, 28, 42, 56, 70 and 84 during Stage 3.
- Placebo: Stage 2 and 3: Placebo matched to IMA-638 subcutaneous injection on Day 1, 8, 28, 42, 56, 70 and 84 during Stage 2 and 3.
Period: Overall Study
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1 | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Started | 16 | 17 | 16 | 16 | 45 | 4 | 45
Completed | 14 | 15 | 16 | 14 | 19 | 0 | 26
Not Completed | 2 | 2 | 0 | 2 | 26 | 4 | 19
Not completed — Adverse Event | 1 | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0 | 3
Not completed — Sponsor's request | 0 | 0 | 0 | 0 | 19 | 4 | 15
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included all randomized participants who received at least 1 dose administration of the test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1 | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3 | Total
Number analyzed (Participants) | 16 | 17 | 16 | 16 | 45 | 4 | 45 | 159
Age, Customized [Number; unit: participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 to 71 years | 16 | 17 | 16 | 16 | 45 | 4 | 45 | 159
  Greater than 71 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 7 | 9 | 25 | 1 | 28 | 91
  Male | 5 | 7 | 9 | 7 | 20 | 3 | 17 | 68

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning (Ante Meridiem) Peak Expiratory Flow Rate (AM PEFR) at Day 112 - Stage 1
Description: The PEFR is a participant's maximum speed of expiration, as measured with a peak flow meter. All participants were issued with the peak flow meter and instructed to perform the activity in triplicate in the morning prior to taking bronchodilator. The best among the 3 readings was selected.
Time Frame: Baseline, Day 112
Population: mITT population (Stage 1) included all randomized participants who received at least 1 dose administration of the test article in Stage 1. Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: liter per minute (L/min)
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 16 | 17 | 16 | 16
liter per minute (L/min)
  Baseline | 286.4 (67.6) | 297.6 (55.4) | 343.5 (91.8) | 291.5 (64.7)
  Change at Day 112 | 21.1 (40.9) | 3.4 (53.6) | 7.6 (38.1) | 11.8 (37.5)

2. Primary Outcome: Change From Baseline in Morning (Ante Meridiem) Peak Expiratory Flow Rate (AM PEFR) at Day 112 - Stage 2/3
Description: as for outcome 1
Time Frame: Baseline, Day 112
Population: mITT population (Stage 2 and 3) included all randomized participants who received at least 1 dose administration of the test article in Stage 2 and 3. LOCF method was used to impute missing values. "n" signifies those participants who were evaluated for this measure at the specified time point for each arm.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 45 | 4 | 45
L/min
  Baseline (n=42, 4, 45) | 329.3 (81.7) | 348.6 (39.9) | 330.4 (89.5)
  Change at Day 112 (n=45, 4, 45) | 6.8 (42.9) | 18.8 (30.7) | 7.6 (48.9)
Statistical Analysis 1: Comparison: IMA-638 200 mg: Stage 2 and 3 vs Placebo: Stage 2 and 3; Day 112: Analysis of co-variance (ANCOVA) model was used with baseline as a covariate, long-acting beta-agonist (LABA) use (Inhaled Corticosteroid [ICS] only or ICS plus LABA) and treatment as two factors; Test type: Superiority or Other; p = 0.612, ANCOVA; Least squares (LS) mean difference = -5.2, 95% CI 2-sided [-25.6 to 15.2]

3. Secondary Outcome: Change From Baseline in Pre-beta-agonist Forced Expiratory Volume in 1 Second (FEV1) at Day 8, 28, 56, 84 and 112 - Stage 1
Description: FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FEV1 was obtained from spirometry, performed before study treatment administration. Participants performed the test in triplicate at each visit and the best of the 3 values was selected.
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: mITT population (Stage 1) included all randomized participants who received at least 1 dose administration of the test article in Stage 1. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 16 | 17 | 16 | 16
liter
  Baseline | 2.1 (0.4) | 2.0 (0.4) | 2.3 (0.5) | 2.0 (0.5)
  Change at Day 8 | 0.1 (0.2) | 0.0 (0.1) | 0.0 (0.3) | -0.0 (0.2)
  Change at Day 28 | 0.1 (0.2) | 0.1 (0.1) | 0.0 (0.4) | 0.0 (0.2)
  Change at Day 56 | 0.0 (0.2) | 0.1 (0.2) | 0.1 (0.3) | 0.1 (0.2)
  Change at Day 84 | 0.1 (0.2) | 0.0 (0.2) | 0.0 (0.4) | 0.1 (0.2)
  Change at Day 112 | 0.2 (0.3) | 0.1 (0.2) | 0.1 (0.4) | 0.1 (0.3)

4. Secondary Outcome: Change From Baseline in Pre-beta-agonist Forced Expiratory Volume in 1 Second (FEV1) at Day 8, 28, 56, 84 and 112 - Stage 2/3
Description: as for outcome 3
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: mITT population (Stage 2 and 3) included all randomized participants who received at least 1 dose administration of the test article in Stage 2 and 3. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 45 | 4 | 45
liter
  Baseline | 2.2 (0.6) | 2.3 (0.7) | 2.1 (0.6)
  Change at Day 8 | -0.0 (0.2) | 0.2 (0.2) | 0.0 (0.3)
  Change at Day 28 | 0.0 (0.3) | 0.2 (0.2) | 0.1 (0.3)
  Change at Day 56 | 0.0 (0.3) | 0.2 (0.2) | 0.1 (0.3)
  Change at Day 84 | 0.1 (0.3) | 0.2 (0.2) | 0.1 (0.3)
  Change at Day 112 | 0.1 (0.3) | 0.2 (0.2) | 0.1 (0.3)
Statistical Analysis 1: Comparison: IMA-638 200 mg: Stage 2 and 3 vs Placebo: Stage 2 and 3; Day 8: ANCOVA model was used with baseline as a covariate, LABA use (ICS only or ICS plus LABA) and treatment as two factors; Test type: Superiority or Other; p = 0.482, ANCOVA; LS mean Difference = -0.0, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 2: Comparison: IMA-638 200 mg: Stage 2 and 3 vs Placebo: Stage 2 and 3; Day 28: ANCOVA model was used with baseline as a covariate, LABA use (ICS only or ICS plus LABA) and treatment as two factors; Test type: Superiority or Other; p = 0.492, ANCOVA; LS mean difference = -0.0, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 3: Comparison: IMA-638 200 mg: Stage 2 and 3 vs Placebo: Stage 2 and 3; Day 56: ANCOVA model was used with baseline as a covariate, LABA use (ICS only or ICS plus LABA) and treatment as two factors; Test type: Superiority or Other; p = 0.323, ANCOVA; LS mean difference = -0.1, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 4: Comparison: IMA-638 200 mg: Stage 2 and 3 vs Placebo: Stage 2 and 3; Day 84: ANCOVA model was used with baseline as a covariate, LABA use (ICS only or ICS plus LABA) and treatment as two factors; Test type: Superiority or Other; p = 0.226, ANCOVA; LS mean difference = -0.1, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 5: Comparison: IMA-638 200 mg: Stage 2 and 3 vs Placebo: Stage 2 and 3; Day 112: ANCOVA model was used with baseline as a covariate, LABA use (ICS only or ICS plus LABA) and treatment as two factors; Test type: Superiority or Other; p = 0.256, ANCOVA; LS mean difference = -0.1, 95% CI 2-sided [-0.2 to 0.1]

5. Secondary Outcome: Change From Baseline in Airway Hyper-reactivity at Day 28 and 112
Description: Airway hyper-reactivity was assessed using provocative concentration 20 (PC20). PC20 was the concentration of methacholine at which participants had 20 percent (%) decrease in FEV1. Results for PC20 were summarized together for all participants who received any dose of IMA-638 and for all participants who received placebo during any stage of the study as per investigator's discretion.
Time Frame: Baseline, Day 28, 112
Population: mITT population included all randomized participants who received at least 1 dose administration of the test article. LOCF method was used to impute missing values. 'N' (Number of Participants Analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: milligram per milliliter (mg/mL)
Groups:
- IMA-638: Included participants who received any dose of IMA-638 subcutaneous injection during Stage 1, 2 or 3.
- Placebo: Included all participants who received placebo matched to IMA-638 subcutaneous injection during Stage 1, 2 or 3.
Arm/Group | IMA-638 | Placebo
Number analyzed (Participants) | 33 | 11
milligram per milliliter (mg/mL)
  Baseline | 1.1 (13.8) | 0.3 (38.9)
  Change at Day 28 | 1.2 (9.8) | 0.6 (11.4)
  Change at Day 112 | 1.0 (28.9) | 0.5 (22.7)
Statistical Analysis 1: Comparison: IMA-638 vs Placebo; Day 28: ANCOVA model was based on the log 2 transformed methacholine challenge test values with baseline as a covariate, LABA use (ICS only or ICS plus LABA) and treatment as two factors; Test type: Superiority or Other; p = 0.090, ANCOVA; LS mean difference = 1.8, 95% CI 2-sided [-0.3 to 3.9]
Statistical Analysis 2: Comparison: IMA-638 vs Placebo; Day 112: ANCOVA model was based on the log 2 transformed methacholine challenge test values with baseline as a covariate, LABA use (ICS only or ICS plus LABA) and treatment as two factors; Test type: Superiority or Other; p = 0.144, ANCOVA; LS mean difference = 2.1, 95% CI 2-sided [-0.8 to 5.0]

6. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-5 (ACQ-5) Score at Day 8, 28, 56, 84 and 112 - Stage 1
Description: ACQ-5 was a 5-item participant-reported questionnaire assessing asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing). Participants were asked to recall how their asthma had been during the previous week. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ score was the mean of the responses. Mean scores of less than or equal to (=<) 0.75 indicate well-controlled asthma, scores between 0.76 and less than (<) 1.5 indicate partly controlled asthma, and a score greater than or equal to (>=) 1.5 indicates uncontrolled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 16 | 17 | 16 | 16
units on a scale
  Baseline | 2.7 (0.6) | 2.6 (0.8) | 2.8 (0.6) | 2.7 (0.7)
  Change at Day 8 | -0.6 (1.1) | -0.2 (0.7) | -0.6 (0.7) | -0.3 (0.6)
  Change at Day 28 | -0.7 (1.1) | -0.5 (0.7) | -0.8 (0.9) | -0.7 (0.6)
  Change at Day 56 | -0.8 (1.1) | -0.6 (0.8) | -1.1 (1.1) | -0.7 (0.7)
  Change at Day 84 | -1.1 (1.2) | -0.8 (0.9) | -1.1 (1.1) | -0.8 (0.8)
  Change at Day 112 | -0.9 (1.2) | -0.7 (0.9) | -1.2 (1.0) | -0.8 (0.8)

7. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-5 (ACQ-5) Score at Day 8, 28, 56, 84 and 112 - Stage 2/3
Description: ACQ-5 was a 5-item participant-reported questionnaire assessing asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing). Participants were asked to recall how their asthma had been during the previous week. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ score was the mean of the responses. Mean scores of =< 0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score >= 1.5 indicates uncontrolled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 45 | 4 | 45
units on a scale
  Baseline | 2.7 (0.6) | 2.3 (0.6) | 2.8 (0.6)
  Change at Day 8 | -0.6 (0.7) | -0.4 (0.8) | -0.5 (0.7)
  Change at Day 28 | -0.7 (1.0) | -0.4 (0.9) | -0.7 (0.8)
  Change at Day 56 | -0.8 (1.1) | -0.4 (0.9) | -0.8 (0.9)
  Change at Day 84 | -0.8 (1.1) | -0.4 (0.9) | -1.0 (0.9)
  Change at Day 112 | -0.8 (1.1) | -0.4 (0.9) | -1.0 (0.9)
Statistical Analysis 1: Comparison: IMA-638 200 mg: Stage 2 and 3 vs Placebo: Stage 2 and 3; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.354, ANCOVA; LS mean difference = -0.1, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 2: Comparison: IMA-638 200 mg: Stage 2 and 3 vs Placebo: Stage 2 and 3; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.900, ANCOVA; LS mean difference = 0.0, 95% CI 2-sided [-0.4 to 0.4]
Statistical Analysis 3: Comparison: IMA-638 200 mg: Stage 2 and 3 vs Placebo: Stage 2 and 3; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.921, ANCOVA; LS mean difference = 0.0, 95% CI 2-sided [-0.4 to 0.4]
Statistical Analysis 4: Comparison: IMA-638 200 mg: Stage 2 and 3 vs Placebo: Stage 2 and 3; [analysis description as in outcome 4, analysis 4]; Test type: Superiority or Other; p = 0.388, ANCOVA; LS mean difference = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 5: Comparison: IMA-638 200 mg: Stage 2 and 3 vs Placebo: Stage 2 and 3; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.249, ANCOVA; LS mean difference = 0.2, 95% CI 2-sided [-0.2 to 0.7]

8. Secondary Outcome: Percentage of Participants Who Required Treatment With Systemic Steroids for Clinical Exacerbation of Asthma - Stage 1
Time Frame: Baseline up to Day 112
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 16 | 17 | 16 | 16
percentage of participants | 0.00 | 0.00 | 6.25 | 12.50
Statistical Analysis 1: Comparison: IMA-638 0.2 mg/kg: Stage 1 vs IMA-638 0.6 mg/kg: Stage 1 vs IMA-638 2 mg/kg: Stage-1 vs Placebo: Stage 1; Test type: Superiority or Other; p = 0.267, Chi-squared

9. Secondary Outcome: Percentage of Participants Who Required Treatment With Systemic Steroids for Clinical Exacerbation of Asthma - Stage 2/3
Time Frame: Baseline up to Day 112
Population: as for outcome 4
Measure: Number; unit: percentage of participant
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 45 | 4 | 45
percentage of participant | 11.11 | 25.00 | 0.00
Statistical Analysis 1: Comparison: IMA-638 200 mg: Stage 2 and 3 vs IMA-638 75 mg: Stage 3 vs Placebo: Stage 2 and 3; Test type: Superiority or Other; p = 0.029, Chi-squared

10. Secondary Outcome: Mean Number of Puffs of Rescue Medication Used - Stage 1
Description: The rescue medication taken for needed symptoms was a short acting beta agonist (SABA) inhaler. Albuterol, 90 microgram (mcg)/puff, was recommended for use.
Time Frame: Day 8, 28, 56, 84, 89, 91, 94, 98, 112
Population: Data for this outcome measure was not analyzed as the study was stopped early and sponsor's decision to analyze only safety and key efficacy outcomes.
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Mean Number of Puffs of Rescue Medication Used - Stage 2/3
Description: The rescue medication taken for needed symptoms was a SABA inhaler. Albuterol, 90 mcg/puff, was recommended for use.
Time Frame: Day 8, 28, 56, 84, 89, 91, 94, 98, 112
Population: as for outcome 10
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Forced Vital Capacity (FVC) - Stage 1
Description: FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: as for outcome 10
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Forced Vital Capacity (FVC) - Stage 2/3
Description: FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: as for outcome 10
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Forced Mid-Expiratory Flow Rate 25 Percent (%) to 75% (FEF25-75) - Stage 1
Description: FEF25-75 is the average expiratory flow over the middle half of the FVC. FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: as for outcome 10
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Forced Mid-Expiratory Flow Rate 25 Percent (%) to 75% (FEF25-75) - Stage 2/3
Description: as for outcome 14
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: as for outcome 10
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Blood Eosinophils Levels - Stage 1
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (cells/L)
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 16 | 17 | 16 | 16
10^9 cells per liter (cells/L)
  Baseline | 0.3 (0.2) | 0.3 (0.2) | 0.3 (0.2) | 0.3 (0.2)
  Day 8 | 0.3 (0.2) | 0.3 (0.2) | 0.3 (0.2) | 0.3 (0.2)
  Day 28 | 0.3 (0.3) | 0.3 (0.4) | 0.3 (0.2) | 0.3 (0.1)
  Day 56 | 0.3 (0.2) | 0.3 (0.3) | 0.3 (0.2) | 0.3 (0.1)
  Day 84 | 0.3 (0.2) | 0.3 (0.3) | 0.3 (0.2) | 0.3 (0.2)
  Day 112 | 0.3 (0.2) | 0.4 (0.3) | 0.3 (0.2) | 0.2 (0.2)

17. Secondary Outcome: Blood Eosinophils Levels - Stage 2/3
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 45 | 4 | 45
10^9 cells/L
  Baseline | 0.3 (0.2) | 0.7 (1.0) | 0.3 (0.2)
  Day 8 | 0.3 (0.2) | 0.7 (1.0) | 0.3 (0.2)
  Day 28 | 0.3 (0.3) | 0.8 (0.9) | 0.3 (0.2)
  Day 56 | 0.3 (0.3) | 0.8 (0.9) | 0.3 (0.1)
  Day 84 | 0.3 (0.3) | 0.8 (0.9) | 0.2 (0.1)
  Day 112 | 0.3 (0.4) | 0.8 (0.9) | 0.2 (0.2)

18. Secondary Outcome: Log 10-transformed Serum Total Immunoglobulin E (IgE) Levels - Stage 1
Description: Log 10-transformed serum total IgE levels were expressed in Log-10 International units/milliliter (IU/mL).
Time Frame: Baseline, Day 28, 56, 84, 112
Population: mITT population (Stage 1) included all randomized participants who received at least 1 dose of test article in Stage 1. LOCF method was used to impute missing values.'N' (Number of Participants Analyzed) signifies participants evaluable for this measure."n" signifies participants evaluated for this measure at the specified time point for each arm.
Measure: Mean (Standard Deviation); unit: log-10 IU/mL
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 16 | 17 | 16 | 16
log-10 IU/mL
  Baseline (n=16, 16, 14, 14) | 3.8 (1.6) | 4.5 (1.9) | 4.4 (1.4) | 4.9 (1.4)
  Day 28 (n=16, 17, 16, 16) | 3.8 (1.5) | 4.3 (1.9) | 4.5 (1.4) | 4.5 (1.7)
  Day 56 (n=16, 17, 16, 16) | 3.7 (1.7) | 4.2 (1.9) | 4.3 (1.5) | 4.6 (1.7)
  Day 84 (n=16, 17, 16, 16) | 3.8 (1.6) | 4.2 (1.9) | 4.4 (1.5) | 4.6 (1.7)
  Day 112 (n=16, 17, 16, 16) | 3.8 (1.6) | 4.1 (1.7) | 4.3 (1.5) | 4.6 (1.7)

19. Secondary Outcome: Log 10-transformed Serum Total Immunoglobulin E (IgE) Levels - Stage 2/3
Description: Log 10-transformed serum total IgE levels were expressed in Log-10 International units/milliliter (IU/mL).
Time Frame: Baseline, Day 28, 56, 84, 112
Population: mITT population (Stage 2 and 3) included all randomized participants who received at least 1 dose administration of the test article in Stage 2 and 3. LOCF method was used to impute missing values. "n" signifies participants evaluated for this measure at the specified time point for each arm.
Measure: Mean (Standard Deviation); unit: log-10 IU/mL
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 45 | 4 | 45
log-10 IU/mL
  Baseline (n=43, 4, 43) | 4.5 (1.5) | 5.1 (1.7) | 4.9 (1.2)
  Day 28 (n=44, 4, 45) | 4.6 (1.5) | 5.1 (1.8) | 4.9 (1.3)
  Day 56 (n=45, 4, 45) | 4.6 (1.5) | 5.1 (1.8) | 4.9 (1.2)
  Day 84 (n=45, 4, 45) | 4.6 (1.5) | 5.1 (1.8) | 4.9 (1.2)
  Day 112 (n=45, 4, 45) | 4.6 (1.5) | 5.1 (1.8) | 5.0 (1.2)

20. Secondary Outcome: Serum Interleukin-13 (IL-13) Level - Stage 1
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: as for outcome 10
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 0 | 0 | 0 | 0

21. Secondary Outcome: Serum Interleukin-13 (IL-13) Level - Stage 2/3
Time Frame: Baseline, Day 8, 28, 56, 84, 112
Population: as for outcome 10
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 0 | 0 | 0

22. Other Pre Specified Outcome: Number of Participants With Vital Sign Abnormalities of Potential Clinical Importance Stage 1
Description: Criteria for potentially clinically important (PCI) vital sign abnormalities- heart rate: greater than (>) 15 beats per minute (bpm) increase from baseline and greater than or equal to (>=) 120 bpm, >15 bpm decrease from baseline and less than or equal to (<=) 45 bpm: systolic blood pressure (SBP): >=20 millimeter of mercury (mmHg) increase from baseline and >=160 mmHg, >=20 mmHg decrease from baseline and <=90 mmHg: diastolic blood pressure (DBP): of >=15 mmHg increase from baseline and >=100 mmHg, >=15 mmHg decrease from baseline and <=50 mmHg, oral temperature <35 or >38.3 degrees centigrade: respiratory rate: <10 or >25 breaths/minute: body weight: >=7% increase or decrease from baseline.
Time Frame: Baseline up to Day 112
Population: mITT population (Stage 1) included all randomized participants who received at least 1 dose administration of the test article in Stage 1.
Measure: Number; unit: participants
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 16 | 17 | 16 | 16
participants | 1 | 2 | 1 | 1

23. Other Pre Specified Outcome: Number of Participants With Vital Sign Abnormalities of Potential Clinical Importance - Stage 2/3
Description: Criteria for PCI vital sign abnormalities- heart rate: >15 bpm increase from baseline and >=120 bpm, >15 bpm decrease from baseline and <=45 bpm: SBP: >=20 mmHg increase from baseline and >=160 mmHg, >=20 mmHg decrease from baseline and <=90 mmHg: DBP: of >=15 mmHg increase from baseline and >=100 mmHg, >=15 mmHg decrease from baseline and <=50 mmHg, oral temperature <35 or >38.3 degrees centigrade: respiratory rate: <10 or >25 breaths/minute: body weight: >=7% increase or decrease from baseline.
Time Frame: Baseline up to Day 112
Population: mITT population (Stage 2 and 3) included all randomized participants who received at least 1 dose administration of the test article in Stage 2 and 3.
Measure: Number; unit: participants
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 45 | 4 | 45
participants | 3 | 0 | 1

24. Other Pre Specified Outcome: Number of Participants With Clinically Important Changes in Physical Findings - Stage 1
Description: Physical examination included examination of general appearance, skin, head, ears, eyes, nose, throat, heart, lungs, breasts, abdomen, external genitalia, extremities, neurological exam, back/spine and lymph nodes.
Time Frame: Baseline up to Day 112
Population: as for outcome 22
Measure: Number; unit: participants
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 16 | 17 | 16 | 16
participants | 0 | 0 | 0 | 0

25. Other Pre Specified Outcome: Number of Participants With Clinically Important Changes in Physical Findings - Stage 2/3
Description: as for outcome 24
Time Frame: Baseline up to Day 112
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 45 | 4 | 45
participants | 0 | 0 | 0

26. Other Pre Specified Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities of Potential Clinical Concern - Stage 1
Description: Clinically significant ECG findings included - heart rate: >15 bpm increase from baseline and >=120 bpm, PR interval: >=20 millisecond (msec) change from baseline and >=220 msec: QRS interval: >=120 msec: corrected QT (QTc) interval: >450 msec for males and >470 msec for females.
Time Frame: Baseline up to Day 112
Population: as for outcome 22
Measure: Number; unit: participants
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 16 | 17 | 16 | 16
participants | 1 | 0 | 1 | 1

27. Other Pre Specified Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities of Potential Clinical Concern - Stage 2/3
Description: Clinically significant ECG findings included - heart rate: >15 bpm increase from baseline and >=120 bpm, PR interval: >=20 msec change from baseline and >=220 msec: QRS interval: >=120 msec: QTc interval: >450 msec for males and >470 msec for females.
Time Frame: Baseline up to Day 112
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 45 | 4 | 45
participants | 3 | 0 | 1

28. Other Pre Specified Outcome: Number of Participants With Injection Site Reaction - Stage 1
Time Frame: Baseline up to Day 112
Population: as for outcome 22
Measure: Number; unit: participants
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 16 | 17 | 16 | 16
participants
  Injection site bruising | 1 | 0 | 0 | 0
  Injection site erythema | 0 | 1 | 0 | 0
  Injection site swelling | 0 | 1 | 0 | 0
  Injection site urticaria | 0 | 1 | 0 | 0

29. Other Pre Specified Outcome: Number of Participants With Injection Site Reaction - Stage 2/3
Time Frame: Baseline up to Day 112
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 45 | 4 | 45
participants
  Injection site bruising | 1 | 0 | 0
  Injection site erythema | 2 | 0 | 1
  Injection site induration | 0 | 0 | 1
  Injection site swelling | 0 | 0 | 1
  Injection site urticaria | 0 | 0 | 1

30. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities of Potential Clinical Importance - Stage 1
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, platelet count, white blood cell count, total neutrophils, eosinophils); hepatobiliary biochemistry: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, total bilirubin, gamma glutamyl transferase (GGT), total lactate dehydrogenase (LDH); renal function tests: blood urea nitrogen (BUN), creatinine, creatinine kinase, uric acid, albumin; electrolytes: sodium, potassium, calcium, magnesium, phosphorus; coagulation: prothrombin time and partial thromboplastin time; glucose: fasting, non-fasting; lipid profile: total cholesterol, triglycerides.
Time Frame: Baseline up to Day 112
Population: as for outcome 22
Measure: Number; unit: participants
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1
Number analyzed (Participants) | 16 | 17 | 16 | 16
participants | 5 | 11 | 12 | 9

31. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities of Potential Clinical Importance - Stage 2/3
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, platelet count, white blood cell count, total neutrophils, eosinophils); hepatobiliary biochemistry: ALT, AST, alkaline phosphatase, total bilirubin, GGT, total LDH; renal function tests: BUN, creatinine, creatinine kinase, uric acid, albumin; electrolytes: sodium, potassium, calcium, magnesium, phosphorus; coagulation: prothrombin time and partial thromboplastin time; glucose: fasting, non-fasting; lipid profile: total cholesterol, triglycerides.
Time Frame: Baseline up to Day 112
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Number analyzed (Participants) | 45 | 4 | 45
participants | 30 | 1 | 21

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | IMA-638 0.2 mg/kg: Stage 1 | IMA-638 0.6 mg/kg: Stage 1 | IMA-638 2 mg/kg: Stage-1 | Placebo: Stage 1 | IMA-638 200 mg: Stage 2 and 3 | IMA-638 75 mg: Stage 3 | Placebo: Stage 2 and 3
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/17 | 2/16 | 1/16 | 2/45 | 0/4 | 0/45
Other Adverse Events (participants affected / at risk) | 13/16 | 12/17 | 11/16 | 10/16 | 27/45 | 1/4 | 26/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMA-638 0.2 mg/kg: Stage 1 (N=16) | IMA-638 0.6 mg/kg: Stage 1 (N=17) | IMA-638 2 mg/kg: Stage-1 (N=16) | Placebo: Stage 1 (N=16) | IMA-638 200 mg: Stage 2 and 3 (N=45) | IMA-638 75 mg: Stage 3 (N=4) | Placebo: Stage 2 and 3 (N=45)
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMA-638 0.2 mg/kg: Stage 1 (N=16) | IMA-638 0.6 mg/kg: Stage 1 (N=17) | IMA-638 2 mg/kg: Stage-1 (N=16) | Placebo: Stage 1 (N=16) | IMA-638 200 mg: Stage 2 and 3 (N=45) | IMA-638 75 mg: Stage 3 (N=4) | Placebo: Stage 2 and 3 (N=45)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tympanic membrane scarring (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual disturbance (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Injection site urticaria (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pitting oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 3
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 0 | 5
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 3 | 13 | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 3 | 1 | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 2 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 4 | 0 | 2
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nicotine dependence (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Pharyngeal leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Diastolic hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was stopped early due to futility of the interim efficacy analysis results. Hence, only safety results and key efficacy results were presented for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.